CLINICAL TRIAL: NCT03611920
Title: Effect of Topical Tetracycline and Dexamethasone on Periodontal and Pulpal Regeneration of Replanted Avulsed Permanent Teeth: A Long-term Follow-up After 9-16 Years
Brief Title: Effect of Topical Tetracycline and Dexamethasone on Periodontal and Pulpal Regeneration of Replanted Avulsed Teeth
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK: 2016-00383
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Dental Trauma; Avulsion; Periodontal Regeneration; Pulpal Regeneration; Topical Dexamethasone; Topical Tetracycline
MeSH Terms: conditions — Fractures, Avulsion | interventions — Tetracycline; Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tetracycline: Teeth were soaked in topical tetracycline 5% for 5 minutes before replantation
  Interventions: Procedure: Tetracycline
- Dexamethasone: Teeth were soaked in dexamethasone (60μ ml-1) for 20 minutes before replantation
  Interventions: Procedure: Dexamethasone

INTERVENTIONS:
Procedure: Tetracycline — Teeth were soaked in topical tetracycline 5% for 5 minutes before replantation
  Groups: Tetracycline
Procedure: Dexamethasone — Teeth were soaked in topical dexamethasone (60μ ml-1) for 20 minutes before replantation
  Groups: Dexamethasone

SUMMARY:
To evaluate the effect of topical tetracycline and dexamethasone on periodontal and pulpal regeneration of avulsed permanent teeth after an observation period between 9-16 years.

DETAILED DESCRIPTION:
Two different medications were applied prior to replantation. A) Topical tetracycline, B) topical dexamethasone. Teeth were splinted using a non-rigid titanium trauma splint for 7-14 days. Endodontic treatment was performed within 1-7 days, except for teeth with an open apex and a short extraoral dry time. All patients received systemic tetracycline for 10 days after accident and were subsequently re-examined.

Follow-up examinations included periodontal examination, percussion, Periotest measurements, pulp sensitivity using CO2 snow, periapical radiograph and intraoral photographs. Additionally a OHIP-14 questionnaire was carried out to determine the oral health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Avulsion of a permanent tooth
* Written informed consent

Exclusion Criteria:

* Extended dry period of more than 60 minutes

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with avulsed permanent teeth who were treated between 2000-2008 at the Department of Oral Surgery, zmk Bern
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2000-08-14 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Number of teeth with periodontal regeneration | After a mean observation period of 12.9±2.4 years (one visit only)
  Periodontal regeneration was assessed with periodontal examination, percussion, Periotest measurements and periapical radiograph.
Number of teeth with pulpal regeneration | After a mean observation period of 12.9±2.4 years (one visit only)
  Pulpal regeneration was assessed with periodontal examination, percussion, Periotest measurements, pulp sensitivity using CO2 snow and periapical radiograph.

SECONDARY OUTCOMES:
Number of teeth that survived | After a mean observation period of 12.9±2.4 years (one visit only)
  Assessed by visual inspection
Number of teeth with open versus closed apex at accident | At baseline
  Assessed by x-ray
Patients satisfaction | After a mean observation period of 12.9±2.4 years (one visit only)
  Measured by OHIP-14 score

CONTACTS AND LOCATIONS:
Overall Officials: Vivianne Chappuis, PD Dr., Study Chair — Department of Oral Surgery and Stomatology, zmk Bern, University Bern
Locations (1):
- zmk Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No